CLINICAL TRIAL: NCT05062837
Title: Hepatectomy Combined With Camrelizumab and Apatinib in CNLC Stage IIIb Hepatocellular Carcinoma
Brief Title: Hepatectomy Combined With Camrelizumab and Apatinib in CNLC Stage IIIb HCC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Guangxi Medical University Cancer Hospital, Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCCA-HCC
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; apatinib

STUDY DESIGN:
Intervention Model Description: Hepatectomy Combined With Camrelizumab and Apatinib
Masking Description: Tumor response will be assessed with revised Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and mRECIST. All imaging data were independently assessed by one radiologist who is blinded to the clinical data and one hepatologist who is not blinded to the clinical data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hepatectomy Combined With Camrelizumab and Apatinib (Experimental): Patients with CNLC IIIb hepatocellular carcinoma will receive hepatectomy. Two to four weeks later, they will receive camrelizumab and apatinib treatments.
  Interventions: Drug: Hepatectomy Combined With Camrelizumab and Apatinib

INTERVENTIONS:
Drug: Hepatectomy Combined With Camrelizumab and Apatinib — Patients with CNLC IIIb hepatocellular carcinoma will receive hepatectomy. Two to four weeks later, they will receive camrelizumab and apatinib treatments.

SUMMARY:
This study intends to prospectively enroll CNLC stage IIIb HCC cases with extrahepatic metastasis and intrahepatic lesions that are expected to be radical resected in several domestic clinical centers, and observe the OS and ORR, DCR, DOR, TTP and PFS of patients receiving hepatectomy combined with apatinib + carrelli pearl treatment.

DETAILED DESCRIPTION:
Carrelizumab was approved by CFDA for second-line indication of hepatocellular carcinoma (HCC) in 2020. The AHELP study led to the CFDA approval of apatinib for second-line indication of HCC in 2021. RESCUE study (phase II) reported the efficacy and safety data of apatinib combined with carrelizumab in first-line (n= 70, 68.6% of CNLC stage IIIb) and second-line (n= 140, 75.8% of CNLC stage IIIb) in the treatment of advanced HCC. ORR was 46% and 25%, 2-year OS was 43% and 45%, median OS was 20.1 and 21.8 months, PFS was 6.4 and 5.5 months, and grade ≥3 adverse events were 78.6% and 76.7%, respectively.

Local progression of intrahepatic lesions of HCC is the most important and direct cause of death, while extrahepatic metastases such as lung and bone metastases progress slowly and pose a much lower threat to life than intrahepatic lesions. For CNLC stage IIIb HCC, although liver resection is not recommended by officical guidelines, for cases with resectable intrahepatic lesions, a number of retrospective studies suggest that patients in the hepatectomy (even palliative resection) group had significantly better OS than those in the nonsurgical group, with a median OS of up to 32 months in the hepatectomy group, significantly higher than 19.2 months in atzuzumab plus bevacizumab or 20.1 months in apatinib plus carrelizumab. Previous retrospective studies in our center also suggest that some HCC patients with extrahepatic metastasis can still benefit from hepatectomy for long-term survival. Other studies suggested that the larger the preoperative diameter of HCC tumor, the greater the probability of postoperative lung metastasis. The more advanced the intrahepatic tumor or the larger the tumor load, the more likely the extrahepatic metastasis. Therefore, hepatectomy combined with targeted drugs +ICI may be the best treatment for HCC with extrahepatic metastasis and radical resection of intrahepatic tumor.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* CNLC stage IIIb HCC with extrahepatic metastasis (such as lymph node, lung, bone metastasis, but not brain metastasis) diagnosed by clinical imaging, and at least one measurable metastasis can be used as RECIST V1.1 to observe the objective efficacy of "targeted + immune" therapy on target lesions;
* Local tumors of the liver are expected to be radically resected;
* Liver function Child-Pugh grade A;
* ICG R15 < 10%;
* ECOG PS 0 or 1 score;
* Estimated survival time ≥6 months;
* Hematological indexes should meet the following conditions: hemoglobin ≥90 g/L; Neutrophil absolute count ≥1.5×109/L; Platelet ≥80×109/L; Total bilirubin ≤1.5×ULN; ALT 3 x ULN or less;AST 3 x ULN or less; Alkaline phosphatase (AKP) ≤2.5×ULN; Serum albumin ≥28 g/L; Serum creatinine ≤1.5×ULN;
* The patient is unwilling to receive TACE or radiotherapy;
* For women of childbearing age, contraceptive measures (such as intrauterine devices, contraceptive tablets or condoms) should be used during the clinical trial until 3 months after the clinical trial ends; Serum or urine HCG test was negative for women of childbearing age within 72 hours prior to study enrollment. Effective contraception should be used during the study period and for three months after the end of the study for male patients with fertile partners.

Exclusion Criteria:

* Have a history or concurrence of other malignancies, except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix;
* Have used or are currently using other immunosuppressive or chemotherapy drugs for HCC (including but not limited to atezolizumab, nivolumab, pembrolizumab, tislelizumab, toripalimab, sintilimab, camrelizumab, S-1, etc.);
* Patients who have received TACE, radiotherapy or systemic therapy within the past 6 months;
* The presence of congenital or acquired immune deficiency diseases (such as HIV positive);
* Known severe allergic reactions to PD-1 mab;
* Within 7 days of enrollment, body temperature of unknown etiology ≥ 38.5℃ or white blood cell count > 15 x 109/L;
* Patients with hemorrhagic diseases (including but not limited to moderate/severe esophagogastric varices, gastrointestinal bleeding, hemorrhagic gastric ulcer, hemoptysis > 2.5 ml per day) within 3 months of enrollment;For cases with positive occult blood in stool, occult blood should be reexamined, and gastroenteroscopy should be performed if necessary);
* Arterial or venous thrombosis, such as cerebrovascular accident (transient ischemic attack, cerebral hemorrhage, cerebral infarction, etc.), deep venous thrombosis and pulmonary infarction, etc., 6 months before enrollment;
* Those who have a history of alcohol or psychotropic drug abuse and cannot get rid of it or have mental disorders;
* Breast-feeding women;
* Autoimmune diseases in active stage or previous autoimmune diseases (such as autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, etc.);
* Were using immunosuppressant or hormone therapy 2 weeks before enrollment;
* Grade 1 CTCAE was not recovered after less than 5 drug half-lives with the last use of molecular targeted therapy or due to adverse events caused by previous therapy;
* Complicated with hepatic encephalopathy or brain metastasis;
* Hypertension beyond drug control (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg);
* Uncontrolled heart disease or symptoms (including but not limited to grade II or higher cardiac function, unstable angina, myocardial infarction in the past 1 year, supraventricular or ventricular arrhythmias requiring treatment or intervention);
* Abnormal coagulation function (INR > 2.0, PT > 16 s), bleeding tendency or need thrombolytic therapy or anticoagulant therapy (but prophylactic use of low-dose aspirin or low-molecular weight heparin is permitted);
* Hereditary or acquired blood diseases (such as hemophilia, thrombocytopenia, coagulation disorders, etc.);
* Urine protein ≥ ++ and 24-hour urine protein ≥ 1.0g in routine urine tests.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  OS is defined as the time from the hepatectomy to death from any cause.

SECONDARY OUTCOMES:
Objective response rate of extrahepatic target lesions | 6 months
  Objective response rate is defined as the proportion of patients with complete response or partial response.

CONTACTS AND LOCATIONS:
Overall Officials: Bang-De Xiang, Ph.D, Principal Investigator — Guangxi Medical University Cancer Hospital
Locations (1):
- Guangxi Medical University Cancer Hospital, Nanning, China

IPD SHARING:
Plan to Share IPD: No
The data underlying this article will be shared on reasonable request to the corresponding author.

REFERENCES:
- [Background] Xu J, Shen J, Gu S, Zhang Y, Wu L, Wu J, Shao G, Zhang Y, Xu L, Yin T, Liu J, Ren Z, Xiong J, Mao X, Zhang L, Yang J, Li L, Chen X, Wang Z, Gu K, Chen X, Pan Z, Ma K, Zhou X, Yu Z, Li E, Yin G, Zhang X, Wang S, Wang Q. Camrelizumab in Combination with Apatinib in Patients with Advanced Hepatocellular Carcinoma (RESCUE): A Nonrandomized, Open-label, Phase II Trial. Clin Cancer Res. 2021 Feb 15;27(4):1003-1011. doi: 10.1158/1078-0432.CCR-20-2571. Epub 2020 Oct 21. PMID 33087333
- [Background] Finn RS, Ikeda M, Zhu AX, Sung MW, Baron AD, Kudo M, Okusaka T, Kobayashi M, Kumada H, Kaneko S, Pracht M, Mamontov K, Meyer T, Kubota T, Dutcus CE, Saito K, Siegel AB, Dubrovsky L, Mody K, Llovet JM. Phase Ib Study of Lenvatinib Plus Pembrolizumab in Patients With Unresectable Hepatocellular Carcinoma. J Clin Oncol. 2020 Sep 10;38(26):2960-2970. doi: 10.1200/JCO.20.00808. Epub 2020 Jul 27. PMID 32716739
- [Background] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160
- [Background] Huang JT, Zhong JH, Zhang J, Gong WF, Ma L, Li LQ, Xiang BD. Hepatectomy combined with apatinib and camrelizumab for CNLC stage IIIb hepatocellular carcinoma: a phase II trial protocol. BMJ Open. 2023 Sep 28;13(9):e067730. doi: 10.1136/bmjopen-2022-067730. PMID 37770273